CLINICAL TRIAL: NCT06391424
Title: Oxygen Consumption (VO2), Effort, and Weaning in the Mechanically Ventilated Patient in the Intensive Care Unit (ICU): EXTUBATE Study
Brief Title: Oxygen Consumption (VO2), Effort, and Weaning in the Mechanically Ventilated Patient in the Intensive Care Unit (ICU)
Acronym: EXTUBATE
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Abraham Schoe, MD, PhD., Intensivist, Department of Intensive Care, Principal Investigator, Associate professor, Leiden University Medical Center
Other Study IDs: P23.068
Record Dates: First submitted 2023-12-15; First posted 2024-04-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Critical Illness; Intensive Care Unit; Oxygen Consumption; Weaning Failure; Mechanical Ventilation; Spontaneous Breathing Trial
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Spontaneous Breathing Trial: Patients who will undergo a spontaneous breathing trial
  Interventions: Diagnostic Test: Spontaneous Breathing Trial

INTERVENTIONS:
Diagnostic Test: Spontaneous Breathing Trial — Patients will undergo an SBT to determine whether they are ready for extubation.

SUMMARY:
In patients who are mechanically ventilated for more than 72 hours weaning failure is a common issue. The Spontaneous breathing trial (SBT) is often done to assess if the patient can be extubated with a high chance of success. However, re-intubation rates are between 15 - 20 % after a successful SBT. The rapid shallow breathing index (RSBI) is an important parameter used in an SBT. Because the high incidence of extubation failure (re-intubation within 48 hours) a search for a better parameter than the RSBI is warranted. Using the measured end-tidal oxygen (etO2) of mechanically ventilated patients it is possible to calculate the VO2, which is a measure of patient effort. The VO2 is a parameter with the potential to predict weaning success or failure, together with other parameters of patient effort like the work of breathing (WOB), pressure time product (PTP) and esophageal pressure swings, reflecting muscle strength of the diaphragm. Therefore, the investigators want to investigate if these parameters are associated with an SBT success or failure.

DETAILED DESCRIPTION:
Weaning failure is a common problem in patients who are mechanically ventilated for more than 72 hours. Prediction of successful extubation is crucial for mechanically ventilated (MV) intensive care patients. Prolonged intubation leads to prolonged mechanical ventilation, which is known to have undesirable and detrimental effects. Premature extubation, on the other hand, is associated with clinical deterioration, a second episode of mechanical ventilation, and prolonged mechanical ventilation, resulting in multiple adverse outcomes.

In addition, up to 20% of all Intensive Care Unit (ICU) patients fail to wean from mechanical ventilation. Prolonged mechanical ventilation is associated with half of the total time spent on the ICU. Improving the prediction of successful weaning provides physicians with a mean to optimize extubation timing, while reducing the incidence of premature extubation.

The rapid shallow breathing index (RSBI) is a parameter commonly used to predict extubation success, next to some other clinical parameters such as consciousness level, the ability to cough and muscle strength. The most commonly used RSBI cut-off value for predicting save extubation incorrectly classifies 15% to 20% of patients. Which means that those patients require another period of mechanical ventilation with possible adverse consequences. It is therefore necessary to develop new parameters or indices aiding in the guidance of extubation timing.

Various other parameters, such as work of breathing (WOB), transpulmonary pressure swings (PS) and the pressure time product (PTP), which are manifestations of patient effort, have been investigated. Although a difference in transpulmonary pressure swings during a spontaneous breathing trial (SBT) has been linked to weaning failure, it has yet to be determined whether transpulmonary pressure swings predict extubation success or failure. For all these measures of effort the placement of an esophageal catheter is obligatory.

Oxygen consumption (VO2) is a direct manifestation of patient effort. It is defined as the difference between the amount of oxygen inhaled and exhaled over a predetermined time interval. Using end tidal oxygen (etO2) measurements and volumetric calculations, it is feasible to track VO2 variations breath-by-breath. A change in oxygen consumption during an SBT could be an early indicator of patient effort and failure.

The investigators hypothesize that VO2 measurement, together with indices of patient effort, could be valuable additional parameters when estimating weaning failure or success, and therefore, aid in the prediction of extubation success or failure.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* > 24 hours mechanically ventilated
* Eligible for a spontaneous breathing trial according to the clinical team
* Regular SBT ("Regulier SBT") according to the Leiden University Medical Center (LUMC) protocol
* Hemodynamically stable
* Esophageal Catheter in situ

Exclusion Criteria:

* Severe chronic obstructive pulmonary disease (COPD) (Gold class IV) if it results in a non regular SBT according to the LUMC protocol.
* Heart failure (LVEF <30%) if it results in a non regular SBT according to the LUMC protocol
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended population consists of adults who are mechanically ventilated in the ICU and meet the criteria for a regular spontaneous breathing trial according to the ruling LUMC protocol.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of weaning failure | 48 hours after SBT
  weaning failure is defined as not meeting the criteria for a succesful spontaneous breathing trial (SBT) or extubation failure, defined as the need for re-intubation within 48 hours, after a succesful SBT and subsequent extubation.
Differences of oxygen consumption during SBT | 10 minutes before, through SBT (average of 30 minutes) and 10 minutes after SBT
  The values of oxygen consumption (in milliliter/minute) and the differences between start, during, and end of the SBT.

SECONDARY OUTCOMES:
Differences of esophageal pressure swings measured with an esophageal catheter during SBT | 10 minutes before, through SBT (average of 30 minutes) and 10 minutes after SBT
  The values of pressure swings (in cmH2O), measured with an esophageal catheter, and the differences between start, during, and end of the SBT.
Differences of work of breathing measured with an esophageal catheter during SBT | 10 minutes before, through SBT (average of 30 minutes) and 10 minutes after SBT
  The values of work of breathing (in Joules/liter), measured with an esophageal catheter, and the differences between start, during, and end of the SBT.
Differences of pressure time product measured with an esophageal catheter during SBT | 10 minutes before, through SBT (average of 30 minutes) and 10 minutes after SBT
  The values of pressure time product (in cmH2O/seconds), measured with an esophageal catheter, and the differences between start, during, and end of the SBT.
Differences of rapid shallow breathing index during SBT | 10 minutes before, through SBT (average of 30 minutes) and 10 minutes after SBT
  The values of rapid shallow breathing index (breaths/minute/liter) and the differences between start, during, and end of the SBT.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Schoe, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Leiden University Medical Centre, Leiden, South Holland
  - Leiden University Medical Center, Leiden

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon request with researchers.

REFERENCES:
- [Background] Trudzinski FC, Neetz B, Bornitz F, Muller M, Weis A, Kronsteiner D, Herth FJF, Sturm N, Gassmann V, Frerk T, Neurohr C, Ghiani A, Joves B, Schneider A, Szecsenyi J, von Schumann S, Meis J. Risk Factors for Prolonged Mechanical Ventilation and Weaning Failure: A Systematic Review. Respiration. 2022;101(10):959-969. doi: 10.1159/000525604. Epub 2022 Aug 17. PMID 35977525
- [Background] Beduneau G, Pham T, Schortgen F, Piquilloud L, Zogheib E, Jonas M, Grelon F, Runge I, Nicolas Terzi, Grange S, Barberet G, Guitard PG, Frat JP, Constan A, Chretien JM, Mancebo J, Mercat A, Richard JM, Brochard L; WIND (Weaning according to a New Definition) Study Group and the REVA (Reseau Europeen de Recherche en Ventilation Artificielle) Network double dagger. Epidemiology of Weaning Outcome according to a New Definition. The WIND Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):772-783. doi: 10.1164/rccm.201602-0320OC. PMID 27626706
- [Background] Epstein SK, Ciubotaru RL, Wong JB. Effect of failed extubation on the outcome of mechanical ventilation. Chest. 1997 Jul;112(1):186-92. doi: 10.1378/chest.112.1.186. PMID 9228375
- [Background] Li F, Nie J, Lu Y, Tong TK, Yi L, Yan H, Fu FH, Ma S. The impact of intermittent exercise in a hypoxic environment on redox status and cardiac troponin release in the serum of well-trained marathon runners. Eur J Appl Physiol. 2016 Oct;116(10):2045-51. doi: 10.1007/s00421-016-3460-5. Epub 2016 Aug 29. PMID 27572505
- [Background] Pham T, Telias I, Beitler JR. Esophageal Manometry. Respir Care. 2020 Jun;65(6):772-792. doi: 10.4187/respcare.07425. PMID 32457170
- [Background] Jubran A, Grant BJ, Laghi F, Parthasarathy S, Tobin MJ. Weaning prediction: esophageal pressure monitoring complements readiness testing. Am J Respir Crit Care Med. 2005 Jun 1;171(11):1252-9. doi: 10.1164/rccm.200503-356OC. Epub 2005 Mar 11. PMID 15764727
- [Background] McClave SA, Kleber MJ, Lowen CC. Indirect calorimetry: can this technology impact patient outcome? Curr Opin Clin Nutr Metab Care. 1999 Jan;2(1):61-7. doi: 10.1097/00075197-199901000-00011. PMID 10453332
- [Background] Takala J, Keinanen O, Vaisanen P, Kari A. Measurement of gas exchange in intensive care: laboratory and clinical validation of a new device. Crit Care Med. 1989 Oct;17(10):1041-7. doi: 10.1097/00003246-198910000-00015. PMID 2676345
- [Background] Bellani G, Foti G, Spagnolli E, Milan M, Zanella A, Greco M, Patroniti N, Pesenti A. Increase of oxygen consumption during a progressive decrease of ventilatory support is lower in patients failing the trial in comparison with those who succeed. Anesthesiology. 2010 Aug;113(2):378-85. doi: 10.1097/ALN.0b013e3181e81050. PMID 20613464
- [Derived] Smits FE, Rietveld PJ, Snoep JWM, van der Velde-Quist F, de Jonge E, Schoe A. P0.1 is an Unreliable Measure of Effort in Support Mechanical Ventilation in Comparison With Esophageal-Derived Measures of Effort: A Comparison Study. Crit Care Med. 2025 Aug 1;53(8):e1650-e1658. doi: 10.1097/CCM.0000000000006745. Epub 2025 Jun 11. PMID 40638487
- [Derived] Smits FE, Rietveld PJ, Snoep JWM, van der Velde-Quist F, de Jonge E, Schoe A. Oxygen consumption, effort, and weaning in the mechanically ventilated patient in the intensive care unit: The extubate study: A protocol for an observational study. Respir Med. 2025 Feb;237:107949. doi: 10.1016/j.rmed.2025.107949. Epub 2025 Jan 16. PMID 39826764